CLINICAL TRIAL: NCT07355023
Title: AI-Enabled Electrocardiogram-Guided Guideline-Directed Medical Therapy on Incident Left Ventricular Dysfunction: A Target Trial Emulation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Ting Liu, Clinical Doctor, Principal Investigator, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202505041
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Left Ventricular (LV) Systolic Dysfunction
Keywords: Artificial intelligence; Electrocardiogram; Deep learning; Left ventricular dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Initiation of Guideline-directed medical therapies, including angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) , beta-blockers and sodium-glucose cotransporter 2 (SGLT2) inhibitors
  Interventions: Behavioral: Guideline-directed medical therapies
- Control (No Intervention): No Guideline-directed medical therapies

INTERVENTIONS:
Behavioral: Guideline-directed medical therapies — Guideline-directed medical therapies for patients at risk of heart failure, including angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) , beta-blockers and sodium-glucose cotransporter 2 (SGLT2) inhibitors.
  Arms: Intervention

SUMMARY:
This multicenter retrospective study evaluates whether artificial intelligence-enabled electrocardiography (AI-ECG) can identify individuals at high risk for left ventricular dysfunction and whether targeted guideline-directed medical therapy can mitigate subsequent risk. Using a large multicenter cohort of patients with preserved left ventricular systolic function, the investigators applied an AI-ECG-based risk stratification approach and emulated a target trial to examine the association between guideline-directed therapies and the risk of incident left ventricular functional decline.

DETAILED DESCRIPTION:
This retrospective, multicenter study utilized electronic medical record (EMR) data from a nationwide healthcare system in Taiwan, comprising one academic medical center and seven regional hospitals. The study period extended from January 2016 through December 2024. Clinical data included demographics, comorbidities, medication prescriptions, 12-lead electrocardiograms, and transthoracic echocardiography results.

An artificial intelligence-enabled electrocardiography (AI-ECG) model was developed to detect left ventricular dysfunction (LVD) using over 50,000 paired ECG-echocardiogram recordings obtained within a 7-day interval. The model architecture consisted of an 82-layer convolutional neural network incorporating an attention mechanism to capture salient temporal and morphological ECG features. The finalized model was applied without modification to the study cohort for risk stratification.

All eligible patients had preserved left ventricular ejection fraction (LVEF) at baseline. Based on AI-ECG predictions at cohort entry, patients classified as having LVD by the model despite normal baseline LVEF were designated as the AI-ECG high-risk group, whereas those predicted not to have LVD were designated as the AI-ECG low-risk group. The primary outcome was incident left ventricular functional decline, defined as a reduction in LVEF to ≤40% on follow-up echocardiography.

Candidate preventive therapies, including angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) , beta-blockers and sodium-glucose cotransporter 2 (SGLT2) inhibitors were first screened by evaluating their individual and combination prescription patterns and their associations with the primary outcome. The most promising therapy identified in this screening phase was subsequently assessed using a target trial emulation framework. Specifically, newly initiated use of the candidate therapy was compared with nonuse to emulate a randomized controlled trial, thereby estimating the effect of early preventive treatment on incident LVEF decline using real-world observational data.

The investigators prespecified analytic methods to estimate causal contrasts using time-to-event analyses suitable for observational data, following emulation of random treatment assignment. Prespecified sensitivity analyses were conducted to assess the robustness of the findings across different clinical settings, comorbidity profiles, concomitant therapies, and alternative AI-ECG risk thresholds.

ELIGIBILITY:
Inclusion Criteria:

* With an ECG followed by an echocardiogram within a 90-day interval
* With preserved left ventricular ejection fraction (LVEF ≥ 50%)

Exclusion Criteria:

* missing essential variables or ECG lead data
* any prior LVEF < 50%
* loss to follow-up or death during the 90-day assessment window

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Rate of left ventricular ejection fraction (LVEF) ≤40% | within follow-up period (up to 10 years)
  Rate of left ventricular ejection fraction (LVEF) ≤40% on follow-up echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No